CLINICAL TRIAL: NCT03187678
Title: A Multicenter, Open-label, Single-sequence Cross-over Study to Assess Safety, Tolerability, and Pharmacokinetics of Intravenous Selexipag in Subjects With Stable Pulmonary Arterial Hypertension Switching From an Oral Stable Dose of Selexipag
Brief Title: Safety Study of the Switch From Oral Selexipag to Intravenous Selexipag in Subjects With Stable Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-065A309; 2016-004035-21 (EudraCT Number)
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: switch; intravenous; selexipag
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selexipag (Experimental): Subjects with stable pulmonary arterial hypertension (PAH) and currently treated with a stable oral dose of Uptravi will be switched to i.v. selexipag from Day 2 to Day 3 (2 infusions on Day 2 and 1 infusion on Day 3). Otherwise, they will continue with their current oral selexipag treatment throughout the study.
  Interventions: Drug: i.v. selexipag; Drug: oral selexipag (Uptravi)

INTERVENTIONS:
Drug: i.v. selexipag — Selexipag for intravenous administration, twice daily as an infusion over 87 min. The dose is individualized for each subject to correspond to his/her current oral dose of Uptravi®.
  Other Names: ACT-293987
Drug: oral selexipag (Uptravi) — Uptravi is used as an auxiliary medicinal product, as part of the PAH standard treatment and administered according to the local prescribing information
  Other Names: ACT-293987

SUMMARY:
The development of selexipag for intravenous administration will be useful to avoid treatment interruptions in patients with pulmonary arterial hypertension (PAH) already treated with selexipag administered orally as tablets (Uptravi®). The target population for intravenous selexipag includes those PAH patients who are hospitalized and are unable to swallow tablets of Uptravi.

The primary objective of this study is to assess whether it is safe for patients with PAH to temporarily change from selexipag tablets (Uptravi®) to selexipag given directly into a vein (intravenous selexipag), and then switching back to the initial oral dose of selexipag.

DETAILED DESCRIPTION:
After screening (Visit 1), each subject will participate in the following consecutive treatment periods: Period 1(treatment with oral selexipag at Visit 2/Day 1), Period 2 (treatment with intravenous selexipag at Visit 2/ Day 2 and Day 3), Period 3 (treatment with oral selexipag starting in the evening of Visit 2/Day 3 and ending 7 to 11 days later at Visit 3). Then a safety follow-up period is planned up to end of study visit (EOS), which occurs between Day 33 and Day 40.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to any study-mandated procedure.
* Male and female subjects aged from 18 to 75 years (inclusive),
* Subjects with stable pulmonary arterial hypertension (PAH) defined as WHO Functional Class I-III at Visit 1 and Visit 2, and no change (i.e., introduction or dose change) in PAH-specific medication (i.e., ERA, PDE-5 inhibitor or sGC stimulator) and diuretics in the last 28 days prior to Visit 2.
* Subjects currently treated with Uptravi® at a stable dose (i.e. unchanged dose) for at least 28 days before Visit 2.
* Women of childbearing potential must have a negative pregnancy test at Visit 1 (screening) and Visit 2.

Exclusion Criteria:

* Pregnant, planning to become pregnant or lactating.
* Known and documented moderate or severe hepatic impairment.
* Subjects having received gemfibrozil at any time since initiation of Uptravi®.
* Treatment with any prostacyclin and prostacyclin analogs within 28 days prior to Visit 1.
* SBP < 90 mmHg at Visit 1 or at Visit 2.
* Known or suspected uncontrolled hyperthyroidism.
* Severe renal failure and ongoing or planned dialysis.
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results.
* Known concomitant life-threatening disease with a life expectancy < 12 months.
* Treatment with another investigational treatment within 3 months of Visit 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Preiss, Study Director — Actelion
Locations (8):
- United States (4):
  - University of California San Diego Medical center - PULM VASCULAR DIV, La Jolla, California
  - TUFTS New England Medical Center - PULM / CRITICAL CARE & SLEEP, Boston, Massachusetts
  - Cleveland Clin Foundation - Dept of Pulm & Critical Care Med, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Germany (4):
  - Universitätsklinikum Giessen und Marburg GmbH, Medizinische Klinik und Poliklinik II, Pneumologie, Giessen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Innere Medizin B, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, II. Medizinische Klinik und Poliklinik, Pneumologie, Hamburg
  - Universitätsklinikum Leipzig / Medizinischen Klinik und Poliklinik I, Pneumologie, Leipzig

REFERENCES:
- [Derived] Klose H, Chin KM, Ewert R, Gall H, Parambil J, Poch D, Seyfarth HJ, Axelsen LN, Hsu Schmitz SF, Stein C, Preston IR. Temporarily switching from oral to intravenous selexipag in patients with pulmonary arterial hypertension: safety, tolerability, and pharmacokinetic results from an open-label, phase III study. Respir Res. 2021 Feb 3;22(1):34. doi: 10.1186/s12931-020-01594-8. PMID 33536021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-two patients treated with Uptravi for pulmonary arterial hypertension (PAH) were screened; 20 of them were enrolled in the study.
Groups:
- Selexipag: Subjects treated with a stable dose of oral selexipag (Uptravi) between 200 and 1600 ug twice daily continued to take Uptravi at their prescribed dose during Period 1 (Day 1), then they were switched to intravenous (iv) selexipag during period 2 (3 doses, Day 2 & Day 3) and back to Uptravi during Period 3
Period: Period 1 (Oral Selexipag)
Arm/Group | Selexipag
Started | 20
Completed | 20
Not Completed | 0
Period: Period 2 (Intravenous Selexipag)
Arm/Group | Selexipag
Started | 20
Completed | 20
Not Completed | 0
Period: Period 3 (Oral Selexipag)
Arm/Group | Selexipag
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or other Pacific Islander | 0
  White | 19
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 13
  United States | 7
World Health Organization Functional classes (WHO FC) [Count of Participants; unit: Participants] — The WHO FC describes the severity of PAH symptoms. It ranges from FC I (no symptoms due to ordinary physical activity) to FC IV (severe symptoms with any activity or at rest). Only PAH patients with WHO FC I, II or III at screening and baseline visits could be enrolled.
  Participants
    FC I | 1
    FC II | 13
    FC III | 6
Uptravi dose at screening [Count of Participants; unit: Participants]
  200 ug twice daily | 0
  400 ug twice daily | 1
  600 ug twice daily | 2
  800 ug twice daily | 2
  1000 ug twice daily | 3
  1200 ug twice daily | 2
  1400 ug twice daily | 1
  1600 ug twice daily | 9
PAH-specific therapies at baseline [Count of Participants; unit: Participants] — The following PAH-specific therapies were allowed on top of Uptravi at baseline: endothelin receptor antagonists (ERA), phosphodiesterase type-5 (PDE5) inhibitors and soluble guanylate cyclase (sGC) stimulators
  Participants
    PDE-5 inhibitors | 1
    sGC stimulator | 1
    ERA + PDE5-inhibitors | 13
    ERA + sGC stimulator | 5
PAH etiology at baseline [Count of Participants; unit: Participants] — Patients with the following types of pulmonary arterial hypertension (PAH) could be enrolled: idiopathic PAH, heritable PAH, PAH associated with another disease or condition, including connective tissue disease (CTD), congenital heart disease (CHD), HIV infection, portal hypertension, schistosomiasis)
  Participants
    Idiopathic PAH | 13
    Heritable PAH | 1
    Drug or toxin induced PAH | 0
    Associated with CTD | 4
    Associated with CHD | 1
    Associated with HIV | 0
    Associated with portal hypertension | 1
    Associated with schistosomiasis | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: AE is any untoward medical event that occurs in a participant during the course of the study whether or not considered by the investigator as related to the study treatment.
Time Frame: From Day 1 to Day 37
Population: Safety analysis set including all enrolled subjects who received at least one dose of Uptravi or intravenous selexipag during any of the study periods
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Participants | 15

2. Primary Outcome: Number of Participants With Prostacyclin-associated Adverse Events
Description: Prostacyclin-associated AE include headache, diarrhea, nausea, vomiting, jaw pain, myalgia, pain in the extremity, flushing and arthralgia.
Time Frame: From Day 1 to Day 37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Participants | 7

3. Primary Outcome: Number of Participants With Adverse Event Related to Injection Site Reactions
Description: This is the number of participants with at least one clinically significant reaction at the injection site (e.g., erythema/redness, tenderness, swelling, induration, hemorrhage at the injection site) occurring on the days of intravenous (iv) selexipag injection.
Time Frame: From Day 2 to Day 3
Population: iv safety analysis set including all enrolled subjects who received at least one dose of intravenous selexipag during Period 2
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Participants | 2

4. Primary Outcome: Number of Participants With Prostacyclin-associated AEs Leading to Study Treatment Discontinuation
Description: This is the number of subjects who discontinued the i.v. selexipag treatment due to prostacyclin-associated adverse events (headache, diarrhea, nausea, vomiting, jaw pain, myalgia, pain in the extremity, flushing and arthralgia).
Time Frame: From Day 2 to Day 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Participants | 0

5. Primary Outcome: Number of Participants With PAH-related Adverse Events
Description: This is the number of participants with at least one AE considered to be related to pulmonary arterial hypertension during the course of the study.
Time Frame: From Day 1 to Day 37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 20
Participants | 3

ADVERSE EVENTS:
Time Frame: From Day 2 to Day 37
Description: Treatment-emergent AEs are reported, i.e. serious and non-serious AEs starting on or after the intravenous injection of selexipag, which is the investigational treatment.
Arm/Group | Selexipag
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=20)
Right Ventricular Failure (Cardiac disorders) | 1 (1)
Blindness Unilateral (Eye disorders) | 1 (1)
Rhegmatogenous Retinal Detachment (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Infusion Site Erythema (General disorders) | 2 (3)
Infusion Site Swelling (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Incorrect Drug Administration Rate (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (9)
Tension Headache (Nervous system disorders) | 1 (2)
Chromaturia (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, Actelion may provide comments and may also request alterations and/or deletions for the sole purpose of protecting its confidential information or patent rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT03187678/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03187678/SAP_001.pdf